CLINICAL TRIAL: NCT05467046
Title: Clinical Relevance of Scratching and Sleep in Atopic Dermatitis
Status: Completed | Type: Observational
Sponsor: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Collaborators: UMC Utrecht (Other)
Responsible Party: Sponsor
Other Study IDs: ICBE-S-000319
Record Dates: First submitted 2022-07-07; First posted 2022-07-20 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Scratching; Sleep
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AD-patients
  Interventions: Device: Smartwatch system

INTERVENTIONS:
Device: Smartwatch system — The Atopic Dermatitis patient cohort is exposed to using a smartwatch system for 5 weeks.

SUMMARY:
Atopic Dermatitis (AD), otherwise known as (atopic) eczema, is a chronic relapsing inflammatory skin disease. For difficult-to-treat AD, treatment options are limited. A better understanding of the underlying immunological cause, led to development of new, targeted therapies. For evaluating effectiveness and making treatment decisions for these new therapies, only 2 subjective methods exist: 1. clinical scores (AD-severity scored by a physician using structured scoring system), 2. questionnaires (completed by AD-patients). Therefore, an objective AD-severity assessment method might provide benefits for clinical practice.

In this study, it is evaluated whether scratching and sleep parameters, obtained with a smartwatch worn by AD-patients, provide added value for clinical practice in dermatology. The usability of this smartwatch system is evaluated by AD-patients.

DETAILED DESCRIPTION:
The study consists of two consecutive parts. In part 1, 30 AD-patient will be asked to wear a smartwatch during nighttime and to complete questionnaires regarding the usability of the smartwatch system. In part 2, a focus group with dermatology Health Care Practitioners (HCPs) will take place. In this focus group, the HCPs will evaluate whether the scratching and sleep parameters obtained from the smartwatches worn by the AD-patients in part 1, provide added value for clinical practice in dermatology.

The primary objective is to collect insights in whether objectification of scratching and sleep in AD-patients during the night provides added value for clinical practice in dermatology. The secondary objective is to collect insights into the requirements of AD-patients and dermatology HCPs for a smartwatch system to be acceptable for use in the dermatology clinical practice.

ELIGIBILITY:
For Atopic Dermatitis patients the eligibility criteria are:

Inclusion Criteria:

* Patient has signed informed consent for the BioDay registry and is enrolled in the BioDay registry.
* Patient has a diagnosis of moderate to severe Atopic Dermatitis, and therefore will be treated with advanced systemic treatment in daily practice according to the Dutch AD guideline (after treatment failure of at least 1 oral immunosuppressive drug or a contra-indication for oral immunosuppressive drugs).
* Patient has no concomitant immunosuppressive therapy at baseline
* Age between 18 and 65 years old (18 years ≤ Age ≤ 65 years).
* Intact skin at both wrists (definition of intact skin: Skin in which there are no breaks, scrapes, cuts, or abnormal openings that allow pathogens to enter).
* Willing and able to provide written informed consent and participate in study procedures.
* Able to understand, read and write Dutch.

Exclusion Criteria:

* Unable to understand instructions
* Expected participation of less than 5 weeks
* Travelling or holiday, for 1 night or more, outside the Netherlands during participation in the study.
* Eczema lesions on one or both wrists at study recruitment
* Patients with neurological disease (e.g., Parkinson's Disease) or physical disability affecting one or both hands, wrist and/or arms.
* Irregular or affected sleep/wake pattern due to causes other than AD. (For example: medical conditions like sleep-apnea or primary insomnia, concomitant medication affecting sleep, alternating shift workers or AD-patients with young infants.)
* Having a tattoo on the upper side of one or both wrists. (Tattoos in the wrist area can cause inaccurate measurements.)
* Institutionalized patients (e.g., care home residents)
* Prisoners (general inmates of prisons or other state institutions)
* Philips research employees
* Study site employees or any other research team member involved directly or indirectly in the conduct of the clinical study
* Cognitively impaired (diagnosis of cognitive impairment in medical file)
* Pregnant persons will not be considered for this study (during pregnancy, the treatment with advanced systemic treatment is not always possible)
* If a patient is not allowed to visit the hospital due to the prevailing COVID-19 restrictions. (If COVID-19 restrictions indicate that it is not allowed to visit the hospital for example when having a positive COVID-19 test, then the patient cannot be included in the study, because it cannot comply with the BioDay study protocol, and thereby indirectly also not with the AD-study protocol).

For dermatology HCPs the eligibility criteria are:

Inclusion criteria

* HCP is allowed to treat AD-patients
* HCP is (trainee) dermatologist, (trainee) physician, (trainee) research-physician, (trainee) nurse practitioner, (trainee) physician assistant or similar, working in the field of dermatology
* HCP has (digitally) signed consent form for the focus group
* HCP works in a hospital that is a member of the BioDay consortium.

Exclusion criteria

* Unable or unwilling to attend focus group
* Philips Research employees

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The atopic dermatitis patients are recruited at the dermatology outpatient clinic of an academic medical center (University Medical Center Utrecht).
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-07 (Actual)

PRIMARY OUTCOMES:
Feedback from dermatology HCPs on whether objectification of nighttime scratching and sleep in AD-patients provides added value for clinical practice in dermatology. | 1 hour, after completion of study part 1

SECONDARY OUTCOMES:
AD-Patient participant feedback via a questionnaire (usability schale) on the acceptability and usability of a wearable-solution for AD-patients. | baseline, and after 5 weeks of participation
Nighttime sleep quality measured with a smartwatch. | baseline, and after 5 weeks of participation
  The following specific sleep quality parameters will be collected, amongst others, Total Sleep Time, Wake After Sleep Onset, Number of Awakenings
Nighttime scratching parameters (e.g., number and duration of scratching periods) determined with a smartwatch. | baseline, and after 5 weeks of participation

CONTACTS AND LOCATIONS:
Overall Officials: Marjolein de Buin-Weller, MD, PhD, Principal Investigator — University Medical Center Utrecht (UMC Utrecht)
Locations (1):
- University of Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No